CLINICAL TRIAL: NCT05776563
Title: Reversibility of Brain Glucose Transport and Metabolism in T2DM
Brief Title: Reversibility of Brain Glucose Transport in Type 2 Diabetes Mellitus (T2DM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000034676; 1K23DK132517-01A1 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aim 1 (Other): Intervention before and after study with subjects with uncontrolled T2DM to measured brain glucose transport specifically in the occipital lobe during acute hyperglycemia
  Interventions: Behavioral: Nutrition visits; Other: Intensification of diabetes regimen; Other: Continuous glucose monitor (CGM)

INTERVENTIONS:
Behavioral: Nutrition visits — Participants will receive exercise and dietary counseling from a nutritionist and registered dietician with extensive experience with diabetes and obesity every 2 weeks during the 12 wee
Other: Intensification of diabetes regimen — Patient will meet every 2 weeks in person or have regular phone calls with an endocrinologist to review glucose control and intensification of the diabetes regimens. Will follow the general strategies outlined in the Position Statement of the American Diabetes Association and the European Association for the Study of Diabetes.
Other: Continuous glucose monitor (CGM) — Individuals with uncontrolled T2DM will be asked use a CGM during the 12 week intervention, to monitor glucose control. Target blood glucose levels will be between 80-130 mg/dl before meals and < 180 mg/dl at bedtime. Individuals not at goal with glycemic targets will undergo intensification of their regimen. Throughout the study, individuals will be contacted via telephone, email or through additional clinic visits as deemed necessary for maintenance of glycemic control.

SUMMARY:
The goal of this clinical trial is to learn about the effects of high blood glucose levels in the brain and assess if the changes seen in individuals with poorly control T2DM can be reversed with good glucose control.

The main question[s] it aims to answer are:

* To determine, whether abnormalities in brain glucose transport seen in individuals with uncontrolled diabetes, can be improved with better glucose control.
* Assess which factors, (duration of diabetes mellitus (DM) and glycemic control) contribute to changes in glucose transport

Participants will have:

* A screening visit
* placement of a continuous glucose monitor (CGM) 2 weeks before the first magnetic resonance spectroscopy (MRS) at week 0
* Additional visits/phone calls for intensification of diabetes management and nutrition visits
* Second magnetic resonance spectroscopy (MRS) at week 12

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-60
* medical history for Type 2 diabetes
* HbA1c > 7.5%, BMI ≥18 kg/m2
* Be willing to adhere to the intensification of their diabetes regimen

Exclusion Criteria:

* Creatinine > 1.5 mg/dL
* Hgb < 10 mg/dL, hematocrit of 37 % for males participants and 33 % for female participants
* ALT >3 x ULN
* untreated thyroid disease,
* uncontrolled hypertension
* known neurological disorders
* untreated psychiatric disorders
* malignancy
* bleeding disorders
* current or recent steroid use in last 3 months
* illicit drug use
* for women: pregnancy, actively seeking pregnancy, or breastfeeding
* inability to enter MRI/MRS (as per standard MRI safety guidelines).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Brain glucose concentration in the occipital cortex week 0 | week 0
  Intracerebral concentrations of glucose across the occipital cortex , as measured by MRS will be compared following hyperglycemic clamp in T2DM individuals at baseline (week0).
Brain glucose concentration in the occipital cortex week 12 | week 12
  Intracerebral concentrations of glucose across the occipital cortex will be compared between T2DM patients before and after 12 weeks of intensification of their diabetes management.

SECONDARY OUTCOMES:
CGM metrics | weeks 12
  Glycemic variability, time above range, time in range and time below range will be assessed by using EasyGV between groups at baseline and after 12 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sanchez Rangel, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital (YNHH) Research Unit (HRU), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No